CLINICAL TRIAL: NCT02112812
Title: A Study on Clinical Response Following Eradication Therapy of Helicobacter Pylori Infection in Parkinson's Disease
Brief Title: Effects of Helicobacter Pylori Infection Eradication in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Dr Norlinah Mohamed Ibrahim, Prof Datin, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF0452012
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Response to Levodopa; Motor Outcomes; Quality of Life Outcomes
Keywords: Parkinsons disease; Helicobacter pylori; Eradication; Levodopa response; Motor outcomes; Quality of Life; Open label
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eradication therapy (Experimental): The patients who were positive for H.pylori infection are entered into an eradication therapy protocol which includes oral esomeprazole 40mg daily, oral clarithromycin 500mg bd and oral amoxicillin 1000mg bd for 14 days.
  Interventions: Drug: Eradication therapy for H.pylori infection; Drug: Eradication of Helcobacter Pylori; Drug: Eradication therapy for Helicobacter pylori

INTERVENTIONS:
Drug: Eradication therapy for H.pylori infection — Patients who were positive for H.pylori infection received an eradication therapy consisting of oral esomeprazole 40 md daily, oral clarithromycin 500mg bd and oral amoxicillin 1000mg bd for 14 days.
Drug: Eradication of Helcobacter Pylori — Patients who are positive on urea breath test are given eradication therapy for 14 days, Eradication therapy includes esomeprazole 40mg daily, clarithromycin 500mg bd, amoxicillin 1g bd
Drug: Eradication therapy for Helicobacter pylori

SUMMARY:
A higher prevalence of Helicobacter pylori infection rate has been demonstrated among PD patients compared to controls. As H. pylori infection is known to interfere with levodopa absorption, we embarked on this is a study to understand the effects of Helicobacter pylori infection eradication among a selected Malaysian population with Parkinsons disease, in relation to levodopa effectiveness and motor improvements.

The study hypotheses are:

1. H. pylori eradication improves L-dopa 'onset' time and prolongs the L-dopa 'on-time' duration.
2. PD patients with H. pylori infection show clinical improvement in motor disability and quality of life after eradication therapy of H. pylori, assessed using UPDRS-III / PDQ39 questionnaires.

DETAILED DESCRIPTION:
Study Background

The earliest observation that there is an association between H. pylori and PD was in 1966 when Strang found that gastric and duodenal ulcers were more common in PD patients than their age and gender-matched controls and that these ulcers preceded the diagnosis of PD by up to 20 years. Upon the discovery of H. pylori and its association with peptic ulcer disease, numerous studies were conducted to look for a correlation between H. pylori and PD.

James Parkinson considered that there may be an association between PD and gastrointestinal pathology when he wrote "Although unable to trace the connection by which a disordered state of the stomach and bowels may induce a morbid action in a part of the medulla spinalis, …little hesitation needs be employed before we determine on the probability of such occurrence" (pg 64, The Shaking Palsy).

A direct causal relationship was hypothesised by Altschuler who proposed that H. pylori might play a part in the biosynthetic route for MPTP or MPTP-like substance that have a direct neurotoxic effect on the dopaminergic neurons.

In 1999, Charlett et al. observed that cardinal features of PD, namely bradykinesia, rigidity and abnormal posture was significantly more prevalent in siblings of PD patients compared to controls. Positive H. pylori serology was found in 70% of PD patients and 63% of their siblings compared to 36-43% of controls. They concluded that familial transmission of H. pylori might account for the significantly higher prevalence of parkinsonism in siblings of PD patients.

Bjarnason et al found that the presence of antibodies against H. pylori correlated with IPD, and eradication showed improvement in the measurement of stride length. There was also a correlation between eradication therapy and reduction in inflammatory markers such as IL-6 and TNF-alpha. They hypothesised that chronic infection leads to underlying chronic inflammatory and autoantibody /molecular mimicry mechanism that leads to destruction of the dopaminergic neurons.

Hirai studied lipid composition of H. pylori and identified three cholesterol glucosidases (CG). Of interest, the similarity of the structure of the CG sterols in H. pylori and sterol glucosidase in cycad, which may hypothesized a possibility that H. pylori with certain strain that can cause parkinsonism by way of producing similar sterol glucosidase that is neurotoxic. Cycad is a type of seed made into flour that has been known to cause ALS-PD disease in population such as in Guam island and Kii,Japan. Murine experimental exposure to cycad showed progressive motor and cognitive deterioration. Pathological analysis revealed that they have loss of motor neurones and loss of striatal dopaminergic terminals.

Levodopa absorption occurs in the duodenum. In advanced PD, gastric motility is impaired and this can delay the transit of levodopa through the pylorus and subsequently, prevent or delay its clinical effect. In the duodenum, any inflammatory pathology can also impair levodopa absorption. H.pylori infection affects L-dopa bioavailability via disruption of duodenal mucosa, the site of its absorption and local production of reactive oxygen species, which may inactivate the drug.

Irregularity in levodopa delivery to the brain is common in PD and can lead to erratic response to levodopa and motor fluctuations. This can be attributed to impaired gastrointestinal transit or absorption of the drug.

Pierantozzi et al. conducted a study in which PD patients with H. pylori infection were randomised into eradication therapy and control groups. Serum levodopa levels were consistently higher in the eradication therapy group compared to controls. The active group was also noted to have prolonged clinical response to levodopa, more "on time" and fewer motor fluctuations.

The authors concluded that H. pylori infection impairs absorption of levodopa and eradication therapy is a simple and inexpensive means to aid levodopa absorption and improve clinical response.

Study justifications

Diagnosing H.pylori infection in Parkinson's patients is important as eradicating H. pylori not only reduces the risk of H. pylori complications such as duodenal ulcer and gastric carcinoma, but it will also help to improve their motor disability. Previous studies abroad have shown that eradication of H. pylori increased levodopa bioavailability as H. pylori had been shown to affect its absorption. Conducting this study among Parkinson's patients in PPUKM will give us data for Malaysian population.

Study Objectives

Primary Objectives:

To compare the clinical response to L-dopa before and after H. pylori eradication therapy in the H. pylori infected PD group. (L-dopa 'onset' time (minutes) and L-dopa 'on-time' duration (minutes) ).

Secondary Objectives:

To assess clinical motor improvement before and after H. pylori eradication therapy in infected PD group, using the UPDRS-III and PDQ39 questionnaires.

Study design and study population. This is a prospective study which, conducted at UKMMC between the months of January 2012 to June 2012. The study population consists of Parkinson's disease patients on levodopa therapy, who will be consecutively recruited from the neurology outpatient clinic UKMMC. The study will be done after the approval of the Research Ethics Committee UKMMC. Patients who fulfill the inclusion and exclusion criteria will be counseled and upon giving informed consent, will be enrolled into the study. Individuals with poor command in English or Bahasa Malaysia will be given explanation with an assistance of an interpreter.

Study protocol and study tools

Upon consent, patients will be enquired regarding their background and the data will be recorded Information regarding sociodemographic characteristics (smoking history, alcohol consumption and coffee consumption), previous antibiotics use, concomitant medical conditions, current medications and any gastrointestinal symptoms will be recorded. Height and weight are measured and recorded into the data collection sheet. The clinical response to L-dopa will be documented (looking at L-dopa 'onset' time (minutes) and L-dopa 'on-time' duration (minutes)). The severity of their Parkinson's disease will be assessed using PDQ-39 questionnaires and the Unified Parkinson's Disease Rating Scale (UPDRS)-III.

Urea Breath test protocol

Each subject undergoes UBT to diagnose H. pylori infection. UBT is selected as the most appropriate tool for diagnosing H. pylori in this study because it is noninvasive, non-radiotoxic and readily available compared to OGDS. Serology testing is cheaper and widely accessible and has been used in many researches locally and internationally. Unfortunately, serology testing has a specificity of 79-90% and sensitivity of 76-84%. Furthermore, patients who are positive for H. pylori will remain seropositive for as long as 4 years after its eradication even when UBT has long been negative.

Subjects who are on PPIs or H2 blockers will be given a later appointment for UBT after 4 weeks of stopping these medications. Each patient will be given 75 mg of IRIS 13C urea mixed in Tang™ Orange juice. Breath sample will be taken at 0 minutes, 10 minutes, 20 minutes and 30 minutes. At each breath, subjects will be asked to inhale deeply and hold for 5 seconds and then blow slowly into a bag until its fully inflated. The breath samples collected will be then analysed using the Non-Dispersive Isotope-Selective InfraRed Spectrometer (NDRIS)[IRIS]. Interpretation of the results are based on the IRIS Software 2.3 for analysis of Delta (δ) over baseline (DOB)

Treatment for H. pylori Patients with positive Urea Breath Test (positive for H. pylori infection) will be started on eradication therapy of H. pylori (oral esomeprazole 40mg twice bd, oral clarithromycin 500mg bd and oral amoxicillin 1000mg bd) for 14 days. This current recommendation was formulated at the Maastricht III Consensus Conference in March 2005.

Follow up visit H pylori-infected Parkinsons disease patients will be followed up in the neurology clinic 3 months after eradication therapy of H pylori. The clinical response to L-dopa after eradication treatment of H pylori will be assessed (looking at L-dopa 'onset' time (minutes) and L-dopa 'on-time' duration (minutes)). The clinical motor improvement will also be assessed using PDQ-39 questionnaires and the Unified Parkinson's Disease Rating Scale (UPDRS)-III. Patients will be guided by investigator to answer the all the questionnaires.

Ethical Consideration

This study will be conducted after the approval of the PPUKM ethics committee. Participants will be explained regarding the procedure and the benefit of the study before they signed the consent form. They are allowed to opt out from the study at any point as they wish.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (PD) by a neurologist
* Age more than 18 years
* Written informed consent given either by the patient or next of kin
* Patient on L-DOPA therapy

Exclusion Criteria:

* Patients with a diagnosis of secondary parkinsonism, and Parkinson's plus syndrome
* History of recent proton pump inhibitors (PPIs) or Histamine (H2) antagonist use for at least 4 weeks prior to the urea breath test
* History of recent antibiotics use (less than 6 months)
* Inability to perform urea breath test

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
1. H. pylori eradication improves L-dopa 'onset' time and prolongs the L-dopa 'on-time' duration. | 3months
  This was measured by asking the patient to determine the time taken to experience on from the time of ingestion of levodopa and to determine the duration of time that they are ON, while receiving levodopa.
  The patients are asked to keep a diary if possible. If not, the patients are asked during their visits, baseline visit, visit 1, visit 2 and visit 3
Improvement in L-dopa 'onset' time and L-dopa 'on-time' duration following H.pylori eradication | 3 months post eradication
  Patients are followed up every 4 weeks, for 12 weeks ( 3 visits). The levodopa onset time is calculated based on the time taken to achieve on following levodopa ingestion, while the ON-time duration is the time the patient remains on following levodopa ingestion.
  Patients are asked to keep a diary, if possible.

SECONDARY OUTCOMES:
Improvement in motor disability after eradication therapy of H. pylori, assessed using UPDRS-III , and improvement in quality of life using PDQ39 | 3 months post eradication
  The patients are followed every 4 weeks, for 3 visits, and their motor disability and quality of life parameters are measured at each visit, while they are ON. The improvement is compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Norlinah Mohamed Ibrahim, MBBCH, MRCP, Principal Investigator — Department of Medicine, Faculty of Medicine, National University of Malaysia
Locations (1):
- UKM Medical Center, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Hashim H, Azmin S, Razlan H, Yahya NW, Tan HJ, Manaf MR, Ibrahim NM. Eradication of Helicobacter pylori infection improves levodopa action, clinical symptoms and quality of life in patients with Parkinson's disease. PLoS One. 2014 Nov 20;9(11):e112330. doi: 10.1371/journal.pone.0112330. eCollection 2014. PMID 25411976